CLINICAL TRIAL: NCT06728111
Title: unRaveling pErioperative MyocArdial INjury
Acronym: REMAIN
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Felix van Lier, Anesthesiologist, Erasmus Medical Center
Other Study IDs: 10945
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Injury; Myocardial Injury After Non-Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High sensitive Troponin T — The baseline population will consist of all patients who underwent a form of non-cardiac surgery. Baseline variables, medication use, type of surgery and perioperative hemodynamic and laboratory variables will be extracted from the hospital information system. One year mortality is registered, as well as major vascular events. This is in line with previous publications from our group. The adjudication strategy used for patients with myocardial injury. For the adjudication process minimal two senior anesthesiologists will be invited. Two members with at least one senior anesthesiologist will receive a sample of patients to adjudicate. Together the entire panel will adjudicate all patients. The goal to investigate the differences between the raters.

SUMMARY:
The aim of this study is to gain insight into the etiology of myocardial injury after non cardiac surgery. Furthermore, suspected etiologies were explored and hierarchically classified into most likely cause how this determines prognosis and what factors are associated with improved outcome.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year of age
* Undergoing non-cardiac surgery in the Erasmus MC, with (high-sensitive) Troponin T > 50 ng/L measured in any of the first three days after surgery.

Exclusion Criteria:

* Re-operations within the study period.
* Daycare surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population to be studied consists of all non-cardiac surgical patients who underwent surgery at Erasmus MC in the period 2017-2023.
Sampling Method: Non-Probability Sample
Enrollment: 1114 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Main etiologies elevated troponin T | from enrollment
  The primary endpoint is a description of the main etiologies found within patients with an elevated troponin T after non cardiac surgery.

SECONDARY OUTCOMES:
Differences in adjudication | from enrollment
  Differences in the adjudication process between different doctors will be assessed according to intraclass coeficients and Fleisch Kappa

CONTACTS AND LOCATIONS:
Overall Officials: Sanne Hoeks, PhD, Study Director — Epidemiologist; Felix van Lier, PhD, Principal Investigator — Anesthesiologist
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT06728111/Prot_000.pdf